CLINICAL TRIAL: NCT01876563
Title: the Effect of Vitamin D on the Serum Thioredoxin, TBP-2, Thioredoxin Reductase, Gene Expression of TBP-2 in Patients With Type II Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17112
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Type 2 Diabetes
Keywords: thioredoxin; TBP-2; thioredoxin reductase; vitamin D; DIABETES
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diabetes, vitamin D (Active Comparator): patients with type 2 diabetes who receive 4000 IU/day vitamin D
  Interventions: Dietary Supplement: vitamin D
- placebo, diabetes (Placebo Comparator): patients with type 2 diabetes who receive one tab placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: vitamin D — one tab 4000 IU/day vitamin D
  Arms: diabetes, vitamin D
Dietary Supplement: placebo — one tab per day placebo
  Arms: placebo, diabetes

SUMMARY:
The aim of this study is the comparision between the effects of vitamin D or placebo supplementation for 2 months in serum level of thioredoxin, TBP-2 and thioredoxin reductase activity in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

literate, willingness to participation, diabetic patients 30- 60 years old, body mass index in the range 18.5- 35, avoidance of dietary supplements, vitamins and herbal products at least 3 months before and throughout the intervention -

Exclusion Criteria:

people who have used vitamin D supplements in last 3 months, having chronic renal disease , GI disease, Hepatobilliary diseases, hematological disorders, hypo- or hyperthyroidism, treatment with orlistat or sibutramine for weight loss, pregnancy and lactation, treatment with insulin or Thiazolidinediones, Smokers

-

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
serum total cholesterol | change from baseline at 2 months
serum HDL cholesterol | change from baseline at 2 months
serum triglycerides level | change from baseline at 2 months
fasting plasma glucose | change from baseline at 2 months
serum LDL cholesterol | change from baseline at 2 months
complete blood count (CBC) | change from baseline at 2 months
HbA1c | change from baseline at 2 months
serum insulin | change from baseline at 2 months
serum calcidiol | change from baseline at 2 months
thioredoxin | change from baseline at 2 months
thioredoxin binding protein 2 (TBP-2) | change from baseline at 2 months
erytrocyte thioredoxin reductase | change from baseline at 2 months

SECONDARY OUTCOMES:
GENE EXPRESSION OF TBP-2 | change from baseline at 2 months

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Tehran University of Medical Sciences, Tehran, Tehran Province
  - Tehran University of Medical Sciences, Tehran